CLINICAL TRIAL: NCT00000636
Title: Prophylaxis Against Tuberculosis (TB) in Patients With Human Immunodeficiency Virus (HIV) Infection and Confirmed Latent Tuberculous Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: CPCRA 004; TB/PPD+; ACTG 177; 11556 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Tuberculosis; Isoniazid; Pyrazinamide; Pyridoxine; Rifampin; AIDS-Related Opportunistic Infections; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Antitubercular Agents; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Tuberculosis; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Isoniazid; Pyrazinamide; Pyridoxine; Rifampin

INTERVENTIONS:
Drug: Isoniazid
Drug: Pyrazinamide
Drug: Pyridoxine hydrochloride
Drug: Rifampin

SUMMARY:
To evaluate and compare the effectiveness of a 2-month regimen of rifampin and pyrazinamide versus a 1-year course of isoniazid (INH) to prevent the development of tuberculosis in patients who are coinfected with HIV and latent Mycobacterium tuberculosis (MTb).

Current guidelines recommend 6 to 12 months of treatment with INH for purified protein derivative (PPD)-positive individuals. Problems with this treatment include compliance, adverse reaction, and the possibility of not preventing disease due to INH-resistant organisms. Studies suggest that two or three months of rifampin and pyrazinamide may be more effective than longer courses of INH. A two-month prevention course should help to increase compliance. In addition, the use of two drugs (rifampin and pyrazinamide) may help overcome problems with drug resistance.

DETAILED DESCRIPTION:
Current guidelines recommend 6 to 12 months of treatment with INH for purified protein derivative (PPD)-positive individuals. Problems with this treatment include compliance, adverse reaction, and the possibility of not preventing disease due to INH-resistant organisms. Studies suggest that two or three months of rifampin and pyrazinamide may be more effective than longer courses of INH. A two-month prevention course should help to increase compliance. In addition, the use of two drugs (rifampin and pyrazinamide) may help overcome problems with drug resistance.

After baseline screening, patients are randomized to one of two treatment arms and are evaluated by means of clinic visits monthly for the first three months, then every three months for the first year (there are additional clinic visits for INH patients). Patients are then evaluated every six months. One group of patients takes INH plus vitamin B6 for 12 months. The other group of patients takes 1 of 2 doses of rifampin (depending on patient's weight) plus pyrazinamide in 3-4 divided doses for 60 days.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral treatment.
* Pneumocystis carinii pneumonia prophylaxis.
* Treatment for acute opportunistic infection/malignancy.
* Aminoglycosides, quinolones or fluoroquinolones such as ciprofloxacin or ofloxacin for < 14 days for treatment of intercurrent infection.

Patients must have:

* HIV infection.
* Signed informed consent.
* Reasonably good health at time of study entry.
* Perceived life expectancy of at least six months.
* Allowed:
* Participation in other clinical trials as long as there is no potential activity of other study drugs against Mycobacterium tuberculosis (MTb), additive toxicities between study agents, or known possible drug interactions between study drugs.

Prior Medication:

Allowed:

* Treatment with quinolones, fluoroquinolones, aminoglycosides, or other agents with known or potential activity against M. tuberculosis.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Current active tuberculosis (confirmed or suspected).
* Sensitivity or intolerance to study medication.
* Acute hepatitis.
* Evidence of peripheral neuropathy, i.e., signs or symptoms of paresis, paresthesias, neuromotor abnormalities, or neurosensory deficits of grade 3 or worse.
* Inability to have concomitant medications changed to avoid serious interaction with study drug.

Concurrent Medication:

Excluded:

-

Quinolones, fluoroquinolones, or aminoglycosides with antituberculous activity (may be used for up to 14 days for treatment of intercurrent infection).Other agents with known or potential antituberculous activity should be avoided, including the following:

* Aminosalicylic acid salts, capreomycin, clofazimine, cycloserine, ethambutol, ethionamide, isoniazid, kanamycin, pyrazinamide, rifabutin, rifampin, streptomycin, and thiacetazone.

Prior Medication:

Excluded:

* History of treatment for > 2 months with agents that have known or potential antituberculous activity other than those specifically allowed.

Agents with potential or known antituberculous activity include the following:

* Aminoglycosides such as amikacin, aminosalicylic acid salts, capreomycin, ciprofloxacin, clofazimine, cycloserine, ethambutol, ethionamide, isoniazid, kanamycin, ofloxacin, pyrazinamide, quinolones or fluoroquinolones, rifabutin, rifampin, streptomycin, and thiacetazone.

Patients may not have:

* Current active tuberculosis.
* Acute hepatitis.
* Peripheral neuropathy of grade 3 or grade 4.

Willing and able, in the clinician's opinion, to comply with the treatment and clinical management issues.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000
Dates: Study Completion 1997-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordin F, Study Chair; Brown LS, Study Chair
Locations (25):
- United States (25):
  - Community Consortium / UCSF, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Hill Health Corp, New Haven, Connecticut
  - Wilmington Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Chicago Dept of Health / Speciality STD Clinic, Chicago, Illinois
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Johns Hopkins Univ / Brazil, Baltimore, Maryland
  - Johns Hopkins Univ / School of Hygiene & Public Health, Baltimore, Maryland
  - Boston Dept of Health and Hosps, Boston, Massachusetts
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - Saint Michael's Med Ctr, Newark, New Jersey
  - Lattimore Comprehensive Pulmonary Disease Clinic, Newark, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Addiction Research and Treatment Corp, Brooklyn, New York
  - Clinical Directors Network of Region II, New York, New York
  - Beth Israel Med Ctr, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Gordin F, Matts J, Miller C, Chaisson R, Garcia M, O'Brien R. Risk factors for developing active tuberculosis (TB) among HIV-infected, PPD-positive (+) patients (pts). Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:151 (abstract no 448)
- [Background] New TB guidelines for persons with HIV. AIDS Treat News. 1998 Nov 6;(No 306):6. PMID 11365963
- [Background] Gordin F, Chaisson RE, Matts JP, Miller C, de Lourdes Garcia M, Hafner R, Valdespino JL, Coberly J, Schechter M, Klukowicz AJ, Barry MA, O'Brien RJ. Rifampin and pyrazinamide vs isoniazid for prevention of tuberculosis in HIV-infected persons: an international randomized trial. Terry Beirn Community Programs for Clinical Research on AIDS, the Adult AIDS Clinical Trials Group, the Pan American Health Organization, and the Centers for Disease Control and Prevention Study Group. JAMA. 2000 Mar 15;283(11):1445-50. doi: 10.1001/jama.283.11.1445. PMID 10732934